CLINICAL TRIAL: NCT02158481
Title: Investigating the Effects of Dietary Ingredients on Vascular Function During Acute Glucose Load
Brief Title: Effects of Dietary Ingredients on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Aspect Clinical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FDS-BNH-0751
Record Dates: First submitted 2014-03-24; First posted 2014-06-06 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Vascular Diseases; Impaired Glucose Tolerance
Keywords: Vascular function; Dietary ingredients; Acute glucose load; Oxidative stress
MeSH Terms: conditions — Vascular Diseases; Glucose Intolerance | interventions — Carotenoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary ingredients: polyphenols and carotenoids (Active Comparator): Dietary ingredients: polyphenols and carotenoids
  Interventions: Dietary Supplement: A capsule containing both polyphenols and carotenoids
- Placebo product (Placebo Comparator): Placebo product
  Interventions: Dietary Supplement: Placebo intervention

INTERVENTIONS:
Dietary Supplement: A capsule containing both polyphenols and carotenoids
  Arms: Dietary ingredients: polyphenols and carotenoids
Dietary Supplement: Placebo intervention — Placebo intervention
  Arms: Placebo product

SUMMARY:
The main aim of the study is to investigate the effects of dietary ingredients (polyphenols and carotenoids) on vascular function during acute glucose load. Each subject will receive 4 weeks of intervention with test product or placebo product after a dietary restriction run-in period of 14 days. Subjects will be challenged with an oral glucose tolerance test (OGTT) immediately after the run-in phase and at the end of the intervention phase. During the OGTT, blood samples will be taken at regular intervals.

The study will be conducted in subjects with impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Males or females confirmed with IGT;
* Age ≥ 35 and ≤ 65 year at screening;
* Body Mass Index (BMI) > 25 and <40 kg/m2;
* Reported intense sporting activities ≤ 10h/w;
* Reported alcohol consumption ≤ 14 units/week (female volunteers) or ≤ 21 units/week (male volunteers)
* Currently not smoking and being a non-smoker for at least six months

Exclusion Criteria:

* Any medical condition or use of over-the-counter and prescribed medication which might affect study measurement (judged by the study physician);
* No reported participation in another nutritional or biomedical trial 3 months before screening;
* Reported weight loss or gain of 10% or more during a period of 6 months prior to screening;
* Anti-hyperglycemic drug or other medication which interferes with study measurements;
* No blood donation 1 month prior to screening;
* Reported allergy or intolerance to test products or other food products provided during the study;

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) levels. | At baseline (after 2 weeks run-in period) and after 4 weeks intervention

SECONDARY OUTCOMES:
Pro-inflammatory and oxidative stress biomarkers | At baseline (after 2 weeks run-in period) and after 4 weeks intervention
  * Luminex HS cytokine, CVD, ADK and MMP panel
  * Endothelial derived factors
  * Systemic inflammatory cytokines: hsTNFα
  * Systemic inflammatory cytokines: hsCRP
  * Endothelial cell function markers
  * Oxidative stress parameters
Cell stress-defence responses | At baseline (after 2 weeks run-in period) and after 4 weeks intervention
  * Direct & indirect markers of cell defence activation
  * Inflammatory and oxidative stress markers
  * Established and exploratory cardiovascular health markers
Clinical chemistry parameters | At baseline (after run-in period of 2 weeks) and after 4 weeks intervention
  * Glucose & Insulin
  * Total cholesterol, LDL, HDL, triglycerides, uric acid, Glycated Serum Proteins & HbA1C.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Thompson, Dr, Principal Investigator — Aspect Clinical
Locations (1):
- Aspect Clinical, Ledbury, United Kingdom